CLINICAL TRIAL: NCT06139120
Title: Evaluation of the Segmental Distribution of Pain Hypersensitivity Among Patients With Central Sensitization Associated With Chronic Subacromial Pain Syndrome
Brief Title: The Segmental Distribution of Hypersensitivity in Patients With Chronic Subacromial Pain Syndrome
Status: Completed | Type: Observational
Sponsor: Cukurova University (Other)
Responsible Party: Principal Investigator, Volkan Deniz, PT, Director, Cukurova University
Other Study IDs: 125/14
Record Dates: First submitted 2023-11-15; First posted 2023-11-18 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Subacromial Pain Syndrome; Central Sensitisation
Keywords: shoulder pain; hypersensitivity; pressure pain threshold
MeSH Terms: conditions — Shoulder Pain; Hypersensitivity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Chronic subacromial pain: Patients with central sensitization associated with chronic pain syndrome
  Interventions: Diagnostic Test: Assessment of hypersensitivity
- Control: Healthy participants
  Interventions: Diagnostic Test: Assessment of hypersensitivity

INTERVENTIONS:
Diagnostic Test: Assessment of hypersensitivity — Assessment of pain hypersensitivity in body segments was performed using pressure pain measurement

SUMMARY:
This study aimed to determine the distribution of pain sensitivity according to body segments in patients with central sensitization associated with chronic subacromial pain syndrome (SPS).This cross-sectional study included patients with chronic SPS and central sensitization (patient group) and the same number of healthy participants as controls. The presence of central sensitization was determined using the Central Sensitization Inventory. To determine the segmental distribution of pain sensitivity, pressure pain threshold measurements were performed bilaterally from the shoulder, forearm, and leg.

DETAILED DESCRIPTION:
Shoulder pain is a common musculoskeletal pain condition in the general population, with a prevalence that has doubled in all age groups over the past 40 years, reaching 22%-30%. Despite treatment, at least 40% of patients report incomplete improvement in pain severity and duration of symptoms, which are the two main determinants of treatment response. There is convincing evidence that the persistence of pain in these patients is due to peripheral or central sensitization mechanisms. Central sensitization refers to pain hypersensitivity mainly resulting from amplifying central nervous system signals and reduced activity of central inhibitory pathways. The clinical presence of central sensitization is determined by examining specific pain characteristics or evaluating changes in pain threshold. The objective manifestation of central sensitization is a decreased pressure-pain threshold (PPT) (hypersensitivity). In previous studies using PPT measurement, pain sensitivity was detected in the shoulder and remote joints in patients with subacromial pain syndrome (SPS), which was considered as evidence of central sensitization. However, these studies did not show how pain sensitivity differs according to body segment in patients with SPS. Hypersensitivity that develops due to chronic shoulder pain would exacerbate the perception of pain caused by other musculoskeletal diseases or trauma. Therefore, it may be important for clinicians to determine how pain sensitivity varies by body segment in patients with SPS

ELIGIBILITY:
Inclusion Criteria:

* To be diagnosed with chronic (≥ 3 months) unilateral SPS according to clinical examination (the Hawkins-Kennedy test and the painful arc test) and/or imaging.
* To be scored ≥ 40 on CSI

Exclusion Criteria:

i) Bilateral shoulder pain syndrome, ii) History ofshoulder surgery, iii) Osteoarthritis of the glenohumeral joint on direct radiography, v)concomitant diseases with the potential risk of development of central/peripheral sensitization [diseases specified in CSI part B, vi) symptomatic lateral/central spinal stenosis, myelopathy, or radiculopathy, vii) history of centrally acting drug use (e.g.,pregabalin, gabapentin, amitriptyline, duloxetine, and opioid) viii) alcohol/substance abuse.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Physical medicine and rehabilitation clinic
Sampling Method: Probability Sample
Enrollment: 116 (Actual)
Dates: Start 2022-09-20 (Actual); Primary Completion 2022-12-20 (Actual); Study Completion 2022-12-30 (Actual)

PRIMARY OUTCOMES:
Pressure pain threshold (PPT) measurement | Baseline
  PPT is the lowest amount of pressure at which pain is felt. The current study used a manual algometer (Force Dial FDK 20, Wagner, Greenwich, USA) with a rubber tip and a surface area of 1 cm2 for PPT measurements. The measurements were performed bilaterally from the shoulder (midpoint of deltoid muscle), forearm (midpoint of brachioradialis muscle), and leg (midpoint of tibialis anterior muscle).
Central sensitization inventory (CSI) | Baseline
  The CSI was used to determine the presence of central sensitization in the participants. The CSI contains 25 items related to central sensitization symptoms scored on a four-point Likert scale, with the total score ranging from 0 to 100. A cutoff score of 40 or greatest indicates the presence of central sensitization.

CONTACTS AND LOCATIONS:
Locations (1):
- Cukurova University, Adana, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No